CLINICAL TRIAL: NCT00283738
Title: A Prospective, Multi-Center, Double-Blinded, Placebo-Controlled Trial to Evaluate the Effectiveness of Patent Foramen Ovale Closure With the BioSTAR Septal Repair Implant to Reduce Refractory Migraine Headache With Aura.
Brief Title: MIST II PFO-Migraine Trial With BioSTAR® Bioabsorbable Septal Repair Implant
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NMT Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: G050119; MIST II
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Migraine; Aura; Patent Foramen Ovale
Keywords: migraine; aura; Patent Foramen Ovale (PFO); cardiac defects; Heart Septal Defects, Atrial; Cephalalgia
MeSH Terms: conditions — Migraine Disorders; Epilepsy; Foramen Ovale, Patent; Heart Septal Defects, Atrial; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Device: BioSTAR Septal Repair Implant System
- 2 (Placebo Comparator): Sham control
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Device: BioSTAR Septal Repair Implant System — PFO Closure
  Arms: 1
Procedure: Sham Procedure — Catheterization
  Arms: 2

SUMMARY:
The objective of the study is to investigate the safety and effectiveness of PFO closure with the BioSTAR Septal Repair Implant System in a population of patients that have refractory migraine (with aura) and who have failed medications.

DETAILED DESCRIPTION:
During the last five years, transcatheter and surgical closure of PFO in the cyrptogenic stroke and TIA population has grown in frequency world-wide. Observational retrospective reports, from both single and multi-center experiences of over 400 patients, suggest Patent Foramen Ovale (PFO) closure to reduce the risk of recurrent migraine events in these populations may be beneficial, particularly for those patients in the migraine with aura subgroup. Although none of these reports are from prospective, randomized, controlled trials, the reports are compelling enough in their totality to support further investigation of a well defined group in a prospective manner. The patients reported in these studies were brought to PFO closure with no expectation of their procedure having any impact on their migraine. In fact, in many cases, the discovery of a history of migraine was not made until well after the PFO closure procedure.

This clinical trial will prospectively compare the safety and effectiveness of PFO closure with the BioSTAR device to a control arm. Patients will be followed one year post-implant.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60.
* migraine history prior to age 50
* must meet definition of refractory migraine with aura
* must have a Patent Foramen Ovale (PFO) within bubble study specifications.
* must provide informed consent. Guardian consent is not accepted.
* patient's heart structure and vasculature must be compatible with BioSTAR Septal Repair Implant System.
* patient must not be pregnant and agrees not to become pregnant during study participation

Exclusion Criteria:

* Medical conditions or medications that are not compatible with protocol or that would increase the patient's risk.
* patient must not have any cardiac or vascular anomalies, repaired or not, that would be incompatible with the delivery system or device for PFO occlusion.
* Currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current trial endpoints.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 610 (Estimated)
Dates: Start 2006-02; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Migraine reduction rates during analysis period.
Safety: Incidence of Major Adverse Cardiac Events (MACE) one year post-implantation.

SECONDARY OUTCOMES:
Efficacy:Change in number of attacks from baseline period compared to analysis phase.
Safety: Device success during index procedure without procedural complication.
Incidence of major AEs during index procedure and post-procedure as they relate to the device and protocol specified medications.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Reisman, MD, Principal Investigator — Swedish Medical Center, Seattle, WA; Stewart J. Tepper, MD, Principal Investigator — Director of the New England Center for Headache
Locations (2):
- United States (2):
  - New England Center for Headache, Stamford, Connecticut
  - Swedish Medical Center, Seattle, Washington